CLINICAL TRIAL: NCT01926639
Title: Radiotherapy Combined With Intratumoral Injections of Dendritic Cells and Rituximab - a Phase II Cancer Vaccine Trial for Patients With Untreated and Relapsed Indolent Non-Hodgkin's Lymphoma
Brief Title: Phase II Cancer Vaccine Trial for Patients With Follicular Lymphoma
Acronym: Lymvac-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Cancer Society (Other); Helse Sor-Ost (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2.2007.1112 Lymvac-1; 2007-002153-23 (EudraCT Number)
Record Dates: First submitted 2013-08-19; First posted 2013-08-21 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Follicular Lymphoma
Keywords: Follicular lymphoma; Rituximab; Autologous dendritic cells; Cancer vaccine
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Radiotherapy; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiotherapy , rituximab and DC (Experimental): Treatment repeated 3 times and targeting different lymph nodes
  Interventions: Biological: Radiotherapy, rituximab and DC

INTERVENTIONS:
Biological: Radiotherapy, rituximab and DC — Lymphoma lymph nodes are irradiated with 8 Gy single treatment and injected with rituximab (5 mg) and autologous DC intratumorally. The treatment is performed 3 times targeting different lymph nodes

SUMMARY:
Patients with non-curable disseminated follicular lymphoma receive local radiotherapy targeting single lymph nodes and injection of low-dose rituximab (anti-CD20) and autologous dendritic cells. The therapy is repeated 3 times, targeting different lesion. Aims are to induce tumor immunity and clinical responses.

DETAILED DESCRIPTION:
The clinical protocol is based on the rationale that the immune system has been developed to combat infectious disease. To mimic the environment in infected tissue, selected tumor-affected lymph nodes are treated locally with a single dose of 8 Gy radiotherapy and injected with therapeutic antibody (anti-CD20/Rituximab). Later, dendritic cells (DC) are injected into the damaged tumor tissue together with a stimulatory cytokine (GM-CSF) to initiate an immune response. Patients with untreated or relapsed stage III/IV follicular lymphoma not in need of standard therapy receive intra-tumoral injections of low-dose anti-CD20 antibodies (5 mg) on days 1 and 3 and local radiotherapy on day 2. On days 4 and 5, dendritic cells generated from monocytes isolated from the patients blood are injected into the site together with the stimulatory cytokine GM-CSF administered subcutaneously. Additional lymph nodes are treated similarly after 2 and 4 weeks. The treatment is thus performed three times, targeting different lymphoma nodes. The primary aims are to induce tumor-specific immune responses and clinical responses.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older
2. Histologically confirmed (by WHO classification) untreated and relapsed indolent non-Hodgkin's B-cell lymphoma of low-grade follicular, marginal zone, lymphoplasmocytic or small lymphocytic subtypes.
3. Stage III/IV
4. Adequate bone marrow function (leukocyte count>2,0, neutrophil count>1.0, platelets>50)
5. Two or more separate lymph nodes > 1,5 cm available for biopsy or treatment.
6. Measurable disease present other than biopsy site and injection site(s).
7. Required wash-out period after previous treatment: Chemotherapy - 8 weeks, Radiotherapy - 4 weeks, Rituximab - 12 weeks
8. WHO status 0-1
9. Life expectancy of more than 6 months
10. Written informed consent
11. Able to comply with the treatment protocol -

Exclusion Criteria:

1. Patients with progressive lymphoma in need of systemic therapy or standard dose irradiation.
2. Chronic bacterial, viral or fungal infection
3. Pre-existing autoimmune or antibody mediated disease including: systemic lupus, erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, autoimmune thrombocytopenia, but excluding controlled thyroid disease, or the presence of autoantibodies without clinical autoimmune disease.
4. Known history of HIV
5. Central nervous system involvement of lymphoma
6. Current anticoagulant therapy which can not safely be paused during treatment injections (ASA < 325 mg/day allowed)
7. Pregnancy -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Response rate | 5 years
  Clinical response measured by CT and PET/CT and immune response

SECONDARY OUTCOMES:
Immune response | 1 year
  Immune response measured by flow cytometry. Peripheral blood mononuclear cells before and after treatment are cultures along with autologous tumor cells. Proliferation is measured.

CONTACTS AND LOCATIONS:
Overall Officials: Arne Kolstad, MD, PhD, Study Chair — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Kolstad A, Kumari S, Walczak M, Madsbu U, Hagtvedt T, Bogsrud TV, Kvalheim G, Holte H, Aurlien E, Delabie J, Tierens A, Olweus J. Sequential intranodal immunotherapy induces antitumor immunity and correlated regression of disseminated follicular lymphoma. Blood. 2015 Jan 1;125(1):82-9. doi: 10.1182/blood-2014-07-592162. Epub 2014 Oct 7. PMID 25293773